CLINICAL TRIAL: NCT04714385
Title: Product Surveillance Registry (PSR) - Targeted Drug Delivery (TDD) - SynchroMed II European Post-Market Clinical Follow-up (PMCF)
Brief Title: Medtronic PSR TDD PMCF
Status: Completed | Type: Observational
Sponsor: Medtronic (Industry)
Responsible Party: Sponsor
Other Study IDs: Medtronic PSR TDD PMCF
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Chronic Pain; Spasticity, Muscle
MeSH Terms: conditions — Chronic Pain; Muscle Spasticity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to provide continuing evaluation and reporting of safety and performance of the SynchroMed II Infusion System within its intended use. Data will support post-market surveillance obligations.

DETAILED DESCRIPTION:
This study was originally posted under NCT01524276 and now posted alone to adapt to new ISO regulation.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legally authorized representative provides written authorization and/or consent per institution and geographical requirements
* Patient has or is intended to receive or be treated with an eligible Medtronic product
* Patient within enrollment window relative to therapy initiation or meets criteria for retrospective enrollment
* The indication for implant meets approved indications
* The patient can reasonably be expected to remain fully on label for a 48-month time period after implant

Exclusion Criteria:

* Patient who is, or will be, inaccessible for follow-up
* Patient with exclusion criteria required by local law
* Patient is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound results
* There is no indication at enrollment (e.g., medical conditions, anticipated relocation, etc.) that the patient will be unable to complete 48 months of follow-up after implant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients implanted with SynchroMed II Model 8637 Programmable Pump who meet approved indications (Chronic pain and severe spasticity)
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Pump accuracy | 4 years
  Demonstrate that the proportion of subjects treated as intended (p) with flow rate accuracy outside the interval of 0.75 to 1.25 (±25 percent) is < 10 percent with 95 percent confidence at 4 years post implant.

SECONDARY OUTCOMES:
Pump survival | 4 years
  Demonstrate pump survival (freedom from product performance events) is > 90 percent at 4 years post-pump implant

CONTACTS AND LOCATIONS:
Locations (15):
- Belgium (5):
  - Brugge, Bruges
  - Leuven, Leuven
  - Roeselare, Roeselare
  - Sint-Niklaas, Sint-Niklaas
  - Wilrijk, Wilrijk
- Praha, Prague, Czechia
- Marseille, Marseille, France
- Netherlands (2):
  - Enschede, Enschede
  - Maastricht, Maastricht
- Ljubljana, Ljubljana, Slovenia
- Spain (2):
  - Badalona, Badalona
  - Madrid, Madrid
- Switzerland (2):
  - Morges, Morges
  - Nottwil, Nottwil
- Middlesbrough, Middlesbrough, United Kingdom